CLINICAL TRIAL: NCT00670787
Title: A Randomized Trial to Establish the Effects of Combination Pill of Losartan Potassium and Hydrochlorothiazide on Medication Compliance Among Patients With High Blood Pressure.
Brief Title: Combination Pill of Losartan Potassium and Hydrochlorothiazide for Improvement of Medication Compliance Trial
Acronym: COMFORT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyushu University (Other)
Responsible Party: Kiyoshi Matsumura, Department of Medicine and Clinical Science, Kyushu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No. 19041
Record Dates: First submitted 2008-04-30; First posted 2008-05-02 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Hypertension
Keywords: Hypertension; combination pill; compliance
MeSH Terms: conditions — Hypertension; Patient Compliance | interventions — Losartan; Hydrochlorothiazide; hydrochlorothiazide, losartan drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combination pill (Active Comparator): Combination pill of losartan potassium 50mg and hydrochlorothiazide 12.5mg in the morning
  Interventions: Drug: Combination pill of losartan and hydrochlorothiazide
- Control group (No Intervention): combination therapy of angiotensin receptor antagonists (losartan potassium 50mg, candesartan 8mg, valsartan 80mg, telmisartan 40mg or olmesartan 20mg) and thiazide or thiazide-like diuretics (hydrochlorothiazide 6.25-12.5mg, trichlormethiazide 0.5-1.0mg, indapamide 0.5-1.0mg or chlorthalidone 6.25-12.5mg)

INTERVENTIONS:
Drug: Combination pill of losartan and hydrochlorothiazide — Combination pill of losartan potassium 50mg and hydrochlorothiazide 12.5mg in the morning
  Other Names: Preminent
  Arms: Combination pill

SUMMARY:
The purpose of the study is to determine whether combination pill of losartan potassium and hydrochlorothiazide will improve medication compliance among patients with high blood pressure.

DETAILED DESCRIPTION:
Despite clear evidence that blood pressure lowering treatment is beneficial for reduction of cardiovascular disease, blood pressure levels are not adequately controlled in many hypertensive patients. More intensive blood pressure lowering treatment is required to achieve maximum reduction of cardiovascular disease. Combination pills of blood pressure lowering drugs could be a safe and effective strategy to achieve blood pressure target but there is no randomized evidence that established the beneficial effects of combination pills of blood pressure lowering drugs. The purpose of the study is to determine whether combination pill of losartan potassium and hydrochlorothiazide will improve medication compliance among patients with high blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 years or above
* Hypertension defined as blood pressure levels of >/=140/90mmHg or current use of blood pressure lowering drugs
* Able to commence combination therapy of angiotensin receptor antagonists and diuretics

Exclusion Criteria:

* Blood pressure measurements of >/=200/120mmHg
* Previous serious adverse events due to angiotensin receptor antagonists or diuretics
* Known or possible pregnancy
* Known severe liver dysfunction
* Known severe kidney disease
* Known contraindication to angiotensin receptor antagonists or diuretics
* Taking >/=4 tablets except for angiotensin receptor antagonists
* ACE inhibitors, thiazide or thiazide-like diuretics in the morning
* Current participation in another clinical trial
* A high likelihood that the patient is not suitable for the study treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2008-06; Primary Completion 2010-11 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Medication compliance | 6 months

SECONDARY OUTCOMES:
Blood pressure | 6 months
cost of blood pressure lowering drugs | 6 months
serious adverse events | 6 months
adverse events | 6 months
blood test | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kiyoshi Matsumura, MD PhD, Principal Investigator — Department of Medicine and Clinical Science, Graduate School of Medical Sciences, Kyushu University
Locations (1):
- Department of Medicine and Clinical Science, Kyushu University, Fukuoka, Fukuoka, Japan